CLINICAL TRIAL: NCT05522803
Title: Can Transcranial Magnetic Stimulation Decrease Food Reinforcement Among Surgical Weight Loss-Seeking Adults Who Have High Levels of Hedonic Hunger and Responsivity to Food Cues
Brief Title: Can Transcranial Magnetic Stimulation Decrease Food Reinforcement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: RHHC20220195
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sequence 1 (Other): TMS followed by sham TMS
  Interventions: Device: TMS followed by sham TMS
- Sequence 2 (Other): Sham TMS followed by TMS
  Interventions: Device: Sham TMS followed by TMS

INTERVENTIONS:
Device: TMS followed by sham TMS — Transcranial Magnetic Stimulation followed by sham TMS
  Arms: Sequence 1
Device: Sham TMS followed by TMS — Sham Transcranial Magnetic Stimulation followed by TMS
  Arms: Sequence 2

SUMMARY:
Reduction in food reinforcement appears to be a principal way by which bariatric surgery lowers energy intake to promote weight loss and other health improvements. However, surgical modulation of mechanisms that influence food reinforcement is variable with some patients appearing more resistant to these effects than others. This "resistant" phenotype, characterized by high levels of hedonic hunger (i.e., eating for pleasure in the absence of hunger) and disinhibition (i.e., susceptibility to cues that promote overeating), can undermine surgical efficacy. Bariatric surgery patients who demonstrate this high-risk eating phenotype may benefit from strategies that can directly target neural mechanisms of food reinforcement. Repetitive transcranial magnetic stimulation (rTMS), a noninvasive procedure that delivers magnetic pulses to stimulate or inhibit nerve cells in the brain, has successfully been used to target dysregulated brain reward circuitry to diminish the reinforcing properties of addictive drugs, such as cocaine. rTMS might have a similar effect on people who have a strong drive to eat in response to the reward of palatable foods. No study has directly examined how rTMS impacts the reinforcing value of food and related brain reward processing among people who find food highly reinforcing. The reinforcing value of food can be measured by comparing how much work a person will choose to do to access that food versus an alternative reinforcer (i.e., relative-reinforcing value of food [RRV]). In this study, we aim to: (1) determine whether rTMS reduces the RRV relative to money; and (2) measure acute rTMS-induced modulation of reward processing with electroencephalography (EEG). Preoperative bariatric patients (n=10) will attend 2 study sessions, at least 1-week apart, with RRV and reward measures completed while EEG is collected before and after a rTMS session. With condition blinding and counterbalancing, participants will be randomized to active rTMS on one day and sham rTMS on the other day. Participants will arrive fasted in the morning, receive a standardized breakfast, complete the RRV and reward tasks during EEG before rTMS (pre-rTMS EEG), receive rTMS, then complete the RRV and reward tasks during EEG after rTMS (post-rTMS EEG). During the active condition, rTMS will be applied to the dorsolateral prefrontal cortex because this region is functionally and structurally connected to the striatum, an area necessary for reward processes. These procedures will allow for comparison of pre- to post-test rTMS changes in behavioral (RRV) and neural modulation (EEG) of food reward between the active and sham conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Seeking to undergo primary (not revisional) bariatric surgery at HH.
2. Be able to give valid informed consent in English.
3. Be 18-60 years of age.
4. Absence of cognitive impairment. Must score below 17 on the adult ADHD self-report scale and have an IQ equivalent of ≥ 80 on the WRAT.
5. Meet clinical criteria regarding hedonic hunger
6. Meet safety criteria for EEG and rTMS.
7. Eat a typical breakfast before 8:00 AM on the day of screening.

Exclusion Criteria:

1. History of any neurological disorder that would increase seizure risk from rTMS such as stroke, brain lesions, previous neurosurgery, any history of seizure or fainting episode of unknown cause, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than one month.
2. First-degree family history of epilepsy, schizophrenia, and bipolar disorder, neurological disorders with a potentially hereditary basis that affect rTMS safety or EEG measures.
3. Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps or sensors, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object in the body that precludes rTMS administration.
4. Noise-induced hearing loss or tinnitus.
5. Current use of any investigational drug or of anti or pro-convulsive action. Use of medications with psychotropic (e.g., benzodiazepines) effects that is not currently stabilized or with disease symptoms present.
6. Lifetime history of schizophrenia, bipolar disorder, mania, or hypomania.
7. History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, and currently under medical care.
8. Participation in any rTMS session less than 2 weeks prior to admission. No rTMS exposure for treatment purposes in the last 6 months.
9. Pregnant women.

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in scores on the Relative-Reinforcing Value (RRV) of Food Questionnaire | The RRV score will be obtained immediately before and immediately after the rTMS and immediately before and after the sham TMS
  Change will be computed as the RRV score after rTMS minus the RRV score before rTMS. RRV will be measured by a validated behavioral choice questionnaire that asks respondents to make a choice between receiving a highly liked food or money. The reinforcing value of food is scored as the choice (1-16) when an individual chooses money instead of food. The higher the number associated with the choice of money, the higher the RRV of food.

CONTACTS AND LOCATIONS:
Overall Officials: Dale Bond, PhD, Principal Investigator — Hartford HealthCare
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bond DS, Papasavas PK, Raynor HA, Grilo CM, Steele VR. Transcranial Magnetic Stimulation for Reducing the Relative Reinforcing Value of Food in Adult Patients With Obesity Pursuing Metabolic and Bariatric Surgery: Protocol for a Pilot, Within-Participants, Sham-Controlled Trial. JMIR Res Protoc. 2023 Nov 6;12:e50714. doi: 10.2196/50714. PMID 37930756